CLINICAL TRIAL: NCT01494558
Title: Phase 3 Study of Etoposide, Cisplatin, and Radiotherapy Versus Paclitaxel, Carboplatin and Radiotherapy in Patients With Unresectable Locally Advanced, Stage III Non-Small Cell Lung Cancer
Brief Title: Study of Etoposide, Cisplatin, and Radiotherapy Versus Paclitaxel, Carboplatin and Radiotherapy to Treat Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Luhua Wang, Chairman of Thoracic Group, Clinical Professor, Radiation Oncology Department, Cancer Hospital&Institute, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006BAI02A02[1]-03
Record Dates: First submitted 2011-12-14; First posted 2011-12-19 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Overall survival
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PE concurrent chemotherapy (Active Comparator): Radiotherapy concurrently with PE chemotherapy
  Interventions: Other: Chemoradiotherapy Regimen between PC and PE
- PC concurrent chemotherapy (Active Comparator): Radiotherapy concurrently with PC chemotherapy
  Interventions: Other: Chemoradiotherapy Regimen between PC and PE

INTERVENTIONS:
Other: Chemoradiotherapy Regimen between PC and PE — etoposide 50mg/m2 d1-5, 29-33 and cisplatin 50mg/m2 d1,8,29 and 36 29-33 during radiotherapy paclitaxel 45mg/m2 weekly and carbplatin AUC =2mg/mL/min weekly during radiotherapy
  Other Names: Chemoradiotherapy

SUMMARY:
Cisplatin-based combination chemotherapy given concurrently with radiotherapy is the standard of care for patients with inoperable stage III NSCLC. The most common chemotherapeutic agents used concurrently with radiotherapy have been vinorelbine, vinblastine, and etoposide in conjunction with cisplatin or weekly paclitaxel and carboplatin. No randomized phase III trials of concurrent chemoradiotherapy have shown the superiority of one chemotherapy regimen over another. The clinical trial is to compare radiotherapy concurrently with PE (etoposide and cisplatin) and PC (paclitaxel and carbplatin) for local advanced NSCLC (stage IIIA/IIIB). It is a randomized, multicenter, open labeled phase III clinical trial. All patients receive conformal radiotherapy or intensity modulated radiotherapy with conventional fraction. The chemotherapy regimens are PE (etoposide 50mg/m2 d1-5, 29-33 and cisplatin 50mg/m2 d1,8,29 and 36 29-33 ) and PC (paclitaxel 45mg/m2 weekly over 1hour and carbplatin AUC =2mg/mL/min over 30min weekly). The primary purpose is to evaluate objective response rate, complications, progression-free survival, overall survival. The second purpose is to evaluate quality of life and cost.

ELIGIBILITY:
Inclusion Criteria:

1. Inoperable stage IIIA/IIIB NSCLC proved by pathology or cytology
2. Age 18 to 75, ECOG ≤ 2, lose weight <10% during 6 months
3. No serious diseases of important organs
4. Chest CT in recently 4 weeks
5. No other tumor disease except stage I cervical cancer or cutaneous basal cell carcinoma
6. Sign consent
7. Measurable lesion

Exclusion Criteria:

1. Pretreatment radiotherapy or chemotherapy
2. Pregnant or lactation woman
3. Serious diseases (include uncontrolled diabetes and infection) of important organs
4. Psychopath
5. Join in other clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-05; Primary Completion 2010-10 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 2 years

SECONDARY OUTCOMES:
Progression Free Survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: luhua Wang, MD, Principal Investigator — Department of Radiation Oncology, Cancer Hospital & Institution, CAMS & PUMC

REFERENCES:
- [Derived] Bi N, Liu L, Liang J, Wu S, Chen M, Lv C, Zhao L, Shi A, Jiang W, Xu Y, Zhou Z, Wang J, Wang W, Chen D, Hui Z, Lv J, Zhang H, Feng Q, Xiao Z, Wang X, Zhang T, Yin W, Li J, He J, Wang L. Efficacy and safety of concurrent chemoradiotherapy in ECOG 2 patients with locally advanced non-small-cell lung cancer: a subgroup analysis of a randomized phase III trial. BMC Cancer. 2020 Apr 6;20(1):278. doi: 10.1186/s12885-020-06780-x. PMID 32252680
- [Derived] Liang J, Bi N, Wu S, Chen M, Lv C, Zhao L, Shi A, Jiang W, Xu Y, Zhou Z, Wang W, Chen D, Hui Z, Lv J, Zhang H, Feng Q, Xiao Z, Wang X, Liu L, Zhang T, Du L, Chen W, Shyr Y, Yin W, Li J, He J, Wang L. Etoposide and cisplatin versus paclitaxel and carboplatin with concurrent thoracic radiotherapy in unresectable stage III non-small cell lung cancer: a multicenter randomized phase III trial. Ann Oncol. 2017 Apr 1;28(4):777-783. doi: 10.1093/annonc/mdx009. PMID 28137739